CLINICAL TRIAL: NCT00261846
Title: A Phase 1/2 Study Of Bosutinib (Ski-606) In Philadelphia Chromosome Positive Leukemias
Brief Title: Study Evaluating SKI-606 (Bosutinib) In Philadelphia Chromosome Positive Leukemias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-200; B1871006, 3160A4-200-WW; 2005-004230-40 (EudraCT Number); B1871006 (Other: Alias Study Number)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Leukemia; tyrosine kinase inhibitor; philadelphia chromosome; Myeloid; Philadelphia Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Philadelphia Chromosome | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SKI-606 (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Part 1, starting dose 400 mg oral, daily dosing in the dose-escalation component.
  Part 2, 500 mg oral, continuous, daily dosing.
  Other Names: SKI-606

SUMMARY:
This is an open-label, continuous daily dosing, two-part safety and efficacy study of SKI-606 (bosutinib) in Philadelphia chromosome positive leukemias (Ph+). Part 1 is a dose-escalation study in chronic phase Chronic Myelogenous Leukemia (CML) subjects to establish the maximum tolerated dose (MTD) in this subject population. Part 2 has begun after the completion of Part 1 and after a dose has been established for the compound in chronic phase subjects. Part 2 is a study of the the efficacy of 500mg daily oral SKI-606 (bosutinib) in patients with all phases of Ph+ CML and Ph+ Acute Lymphocytic Leukemia (ALL). The protocol will test the hypotheses that oral daily dosing of bosutinib at 500 mg will attain (1) Major Cytogenetic Response (MCyR) in chronic phase CML patients and (2) Overall Hematological Response (OHR) in advanced leukemia patients. Each phase of the disease will be evaluated as a separate cohort.

ELIGIBILITY:
Inclusion Criteria:

* Ph+ CML or Ph+ ALL who are primarily refractory to full-dose imatinib (600 mg), have disease progression/relapse while on full-dose imatinib, or are intolerant of any dose of imatinib.
* At least 3 months post stem cell transplantation
* Able to take daily oral capsules/tablets reliably

Exclusion Criteria:

* Subjects with Philadelphia chromosome, and bcr-abl negative CML
* Overt leptomeningeal leukemia
* Subjects without evidence of leukemia in bone marrow (extramedullary disease only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2006-01-18 (Actual); Primary Completion 2009-09-25 (Actual); Study Completion 2015-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (110):
- United States (28):
  - City of Hope National Medical Center, Duarte, California
  - HealthONE Presbyterian, Denver, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Oncology Specialists, S.C., Niles, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - University Of Maryland Medical Center, Baltimore, Maryland
  - University Of Maryland, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hudson Valley Hematology and Oncology Associates, Hawthorne, New York
  - Westchester Oncology Hematology Group, P.C., Hawthorne, New York
  - Westchester Oncology Hematology, Group, P.C., Hawthorne, New York
  - New York Presbyterian Hospital, New York, New York
  - University of Rochester Cancer Center Pharmacy, Rochester, New York
  - University of Rochester Medical Center Strong Memorial Hospital - James P. Wilmot Cancer Center, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Rochester-James P. Wilmot Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Westchester Medical Center, Valhalla, New York
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (8):
  - Hospital universitario austral, Pcia de Buenos Aires, Argentina
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Hospital Britanico, Buenos Aires
  - Academia Nacional de Medicina-Instituto de Investigaciones Hematologicas, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Clinica del Sol, Buenos Aires
  - Centro Medico S.A., Corrientes
  - Hospital Jose Ramon Vidal, Corrientes
- Australia (5):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Institute of Medical and Veterinary Science, Adelaide
  - Department of Clinical Haematology and Bone Marrow Transplantation, Melbourne
  - Royal Brisbane and Women's Hospital, Queensland
  - Haematology and Oncology Clinics of Australia, Queensland
- Klinikum Kreuzschwestern Wels, Wels, Austria
- Brazil (4):
  - Hospital Brigadeiro da Secretaria de Estado da Saude de Sao Paulo, Jardim Paulista, Sao Paulo/sp - Brazil
  - Centro de Estudos da Disciplina dr Hematologia da Faculdade de Medicine do ABC, Santo André, Sp - Brazil
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Sp Brazil
  - Hospital de Clinicas - Universidade Federal do Parana, Curitiba, PR
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis, Jewish General Hospital, Montreal, Quebec
- Instituto Clinico Oncologico del Sur, Temuco, Chile
- China (5):
  - The First Hospital affiliated to the Medical School of Zhejiang University, Zhejiang, P.r China
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing, P.r. China
  - The Department of Hematology, The Chinese PLA General Hospital, Beijing, P.r. China
  - The Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, P.r. China
  - The Department of Hematology, Ruijin Hospital Affiliated to School of Medicine of Shanghai Jiaotong, Shanghai
- Colombia (2):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Fundacion Santa Fe de Bogota, Bogota, Cundinamarca
- Biomedicum Helsinki, Helsinki, Finland
- Germany (10):
  - Universitaet Mainz, Mainz, Rhineland-Palatinate
  - University Hospital Carl Gustav Carus, Dresden
  - Universitaetsklinikum Hamburg - Eppendorf, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Magdeburg A. oe. R., Magdeburg
  - III Medizinische Klinik und Poliklinik, Mainz
  - Klinikum der Johann Gutenberg Universitaet Mainz, Mainz
  - Universitaet Mainz Iii. Medizinische Klinik Abteilung Fuer Haematologie, Mainz
  - Universitaetsklinikum Mainz, Mainz
  - III. Medizinische Klinik, Mannheim
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hosp., Chai Wan
  - Queen Mary Hospital, Hong Kong
- Fovarosi Onkormanyzat Egyesitett Szent Istvan es Szent Laszlo, Budapest, Hungary
- Christian Medical College, Vellore, Tamil Nadu, India
- Italy (4):
  - University of Bologna, Bologna, Province of Bologna
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano, Torino
  - AOU-S.Orsola-Malpighi - Universita degli Studi di Bologna, Bologna
  - Azienda Ospedaliera San Gerardo, Monza
- Mexico (2):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Nuevo León
  - Centro Oncologico Estatal ISSEMYM, Toluca Estado de Mexico
- Netherlands (5):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - UMCG - Pharmacy, Groningen
  - Universitair Medisch Centrum Groningen, Groningen
  - VUMC, The Netherlands
- Avd. for blodsykdommer, Trondheim, Norge, Norway
- Hospital Nacional Edgardo Rebagliati Martins, Lima, Peru
- Russia (6):
  - Kirov Research Institute of Hematology and Blood transfusion of Roszdrav Hematology clinic, Kirov
  - Hematological Research Centre of RAMS, Moscow
  - Moscow regional Clinical Research Institute named after M.F Vladimirsky, Moscow
  - Rostov State Medical University of Roszdrav, Rostov-on-Don
  - Saint Petersburg State Medical University Hematology Department, Saint Petersburg
  - State Healthcare Institution, Sverdlovsk Regional Clinical Hospital, Yekaterinburg
- Singapore General Hospital, Singapore, Singapore
- South Africa (4):
  - University of the Free State, Bloemfontein
  - University of Cape Town, Cape Town
  - Johannesburg Hospital, Parktown
  - Clinical Haematology Unit, Soweto
- South Korea (2):
  - The Catholic University of Korea, Seoul St. Mary Hospital, Seoul
  - Dept. of Hematology, Seoul
- Spain (4):
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona, Catalonia
  - Hospital Universitari Clinic de Barcelona, Barcelona, Catalonia
  - Hospital Universitario La Princesa, Madrid
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
- Akademiska University Hospital, Uppsala, Sweden
- National Taiwan University Hospital - Section of Hematology-Oncology, Taipei, Taiwan
- United Kingdom (4):
  - Northern Centre for Cancer Care - The Newcastle Upon Tyne Hospitals - NHS Foundation Trust, Newcastle upon Tyne, North East England
  - School of Clinical and Laboratory Sciences, University Upon Tyne, North East England
  - Hammersmith Hospital, London
  - Clinical Research Facility, Newcastle Upon Tyne, North East England

REFERENCES:
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Kota V, Brummendorf TH, Gambacorti-Passerini C, Lipton JH, Kim DW, An F, Leip E, Crescenzo RJ, Ferdinand R, Cortes JE. Efficacy and safety following bosutinib dose reduction in patients with Philadelphia chromosome-positive leukemias. Leuk Res. 2021 Dec;111:106690. doi: 10.1016/j.leukres.2021.106690. Epub 2021 Aug 21. PMID 34673442
- [Derived] Gambacorti-Passerini C, Cortes JE, Lipton JH, Kantarjian HM, Kim DW, Schafhausen P, Crescenzo R, Bardy-Bouxin N, Shapiro M, Noonan K, Leip E, DeAnnuntis L, Brummendorf TH, Khoury HJ. Safety and efficacy of second-line bosutinib for chronic phase chronic myeloid leukemia over a five-year period: final results of a phase I/II study. Haematologica. 2018 Aug;103(8):1298-1307. doi: 10.3324/haematol.2017.171249. Epub 2018 May 17. PMID 29773593
- [Derived] Kantarjian HM, Mamolo CM, Gambacorti-Passerini C, Cortes JE, Brummendorf TH, Su Y, Reisman AL, Shapiro M, Lipton JH. Long-term patient-reported outcomes from an open-label safety and efficacy study of bosutinib in Philadelphia chromosome-positive chronic myeloid leukemia patients resistant or intolerant to prior therapy. Cancer. 2018 Feb 1;124(3):587-595. doi: 10.1002/cncr.31082. Epub 2017 Oct 26. PMID 29072772
- [Derived] Cortes JE, Khoury HJ, Kantarjian HM, Lipton JH, Kim DW, Schafhausen P, Matczak E, Leip E, Noonan K, Brummendorf TH, Gambacorti-Passerini C. Long-term bosutinib for chronic phase chronic myeloid leukemia after failure of imatinib plus dasatinib and/or nilotinib. Am J Hematol. 2016 Dec;91(12):1206-1214. doi: 10.1002/ajh.24536. Epub 2016 Sep 15. PMID 27531525
- [Derived] Whiteley J, Reisman A, Shapiro M, Cortes J, Cella D. Health-related quality of life during bosutinib (SKI-606) therapy in patients with advanced chronic myeloid leukemia after imatinib failure. Curr Med Res Opin. 2016 Aug;32(8):1325-34. doi: 10.1185/03007995.2016.1174108. Epub 2016 May 5. PMID 27045164
- [Derived] Hsyu PH, Mould DR, Abbas R, Amantea M. Population pharmacokinetic and pharmacodynamic analysis of bosutinib. Drug Metab Pharmacokinet. 2014;29(6):441-8. doi: 10.2133/dmpk.DMPK-13-RG-126. Epub 2014 Jun 10. PMID 24919837 (Retraction: PMID 30922682 Drug Metab Pharmacokinet. 2019 Apr;34(2):163)
- [Derived] Gambacorti-Passerini C, Brummendorf TH, Kim DW, Turkina AG, Masszi T, Assouline S, Durrant S, Kantarjian HM, Khoury HJ, Zaritskey A, Shen ZX, Jin J, Vellenga E, Pasquini R, Mathews V, Cervantes F, Besson N, Turnbull K, Leip E, Kelly V, Cortes JE. Bosutinib efficacy and safety in chronic phase chronic myeloid leukemia after imatinib resistance or intolerance: Minimum 24-month follow-up. Am J Hematol. 2014 Jul;89(7):732-42. doi: 10.1002/ajh.23728. Epub 2014 Apr 28. PMID 24711212
- [Derived] Kantarjian HM, Cortes JE, Kim DW, Khoury HJ, Brummendorf TH, Porkka K, Martinelli G, Durrant S, Leip E, Kelly V, Turnbull K, Besson N, Gambacorti-Passerini C. Bosutinib safety and management of toxicity in leukemia patients with resistance or intolerance to imatinib and other tyrosine kinase inhibitors. Blood. 2014 Feb 27;123(9):1309-18. doi: 10.1182/blood-2013-07-513937. Epub 2013 Dec 17. PMID 24345751
- [Derived] Trask PC, Cella D, Powell C, Reisman A, Whiteley J, Kelly V. Health-related quality of life in chronic myeloid leukemia. Leuk Res. 2013 Jan;37(1):9-13. doi: 10.1016/j.leukres.2012.09.013. Epub 2012 Oct 29. PMID 23116602
- [Derived] Khoury HJ, Cortes JE, Kantarjian HM, Gambacorti-Passerini C, Baccarani M, Kim DW, Zaritskey A, Countouriotis A, Besson N, Leip E, Kelly V, Brummendorf TH. Bosutinib is active in chronic phase chronic myeloid leukemia after imatinib and dasatinib and/or nilotinib therapy failure. Blood. 2012 Apr 12;119(15):3403-12. doi: 10.1182/blood-2011-11-390120. Epub 2012 Feb 27. PMID 22371878
- [Derived] Trask PC, Cella D, Besson N, Kelly V, Masszi T, Kim DW. Health-related quality of life of bosutinib (SKI-606) in imatinib-resistant or imatinib-intolerant chronic phase chronic myeloid leukemia. Leuk Res. 2012 Apr;36(4):438-42. doi: 10.1016/j.leukres.2011.10.011. Epub 2011 Oct 28. PMID 22036634
- [Derived] Cortes JE, Kantarjian HM, Brummendorf TH, Kim DW, Turkina AG, Shen ZX, Pasquini R, Khoury HJ, Arkin S, Volkert A, Besson N, Abbas R, Wang J, Leip E, Gambacorti-Passerini C. Safety and efficacy of bosutinib (SKI-606) in chronic phase Philadelphia chromosome-positive chronic myeloid leukemia patients with resistance or intolerance to imatinib. Blood. 2011 Oct 27;118(17):4567-76. doi: 10.1182/blood-2011-05-355594. Epub 2011 Aug 24. PMID 21865346
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A4-200&StudyName=Study%20Evaluating%20SKI-606%20%28Bosutinib%29%20In%20Philadelphia%20Chromosome%20Positive%20Leukemias

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib 400 mg (Part 1): Single oral dose of bosutinib 400 milligram (mg) on Day 1 and then bosutinib 400 mg orally once daily continuously from Day 3 up to Week 4. All participants who completed treatment in Part 1 were continued in chronic phase second-line (CP2L) chronic myelogenous leukemia (CML) Part 2 of the study.
- Bosutinib 500 mg (Part 1): Single oral dose of bosutinib 500 mg on Day 1 and then bosutinib 500 mg orally once daily continuously from Day 3 up to Week 4. All participants who completed treatment in Part 1 were continued in CP2L-CML Part 2 of the study.
- Bosutinib 600 mg (Part 1): Single oral dose of bosutinib 600 mg on Day 1 and then bosutinib 600 mg orally once daily continuously from Day 3 up to Week 4. Eleven participants who completed treatment in Part 1 were continued in CP2L-CML Part 2 of the study and 1 participant was continued in advanced phase (AP) CML Part 2 of the study.
- Bosutinib 500 mg, CP2L-CML IM-R (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP2L IM-R CML; who had no prior proto-oncogene tyrosine-protein kinase Src, Abl, or Src-Abl inhibitor exposure other than IM.
- Bosutinib 500 mg, CP2L-CML IM-I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP2L IM-I CML; who had no prior proto-oncogene tyrosine-protein kinase Src, Abl, or Src-Abl inhibitor exposure other than IM.
- Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP3L IM R/I, D and NI R/I or IM R/I and NI-I CML.
- Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP3L IM R/I and D-R CML.
- Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP3L IM R/I and D-I CML.
- Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with CP3L IM R/I and NI-R CML.
- AP-CML Total (Part 2): All participants who received bosutinib 500 mg orally once daily in AP CML who were IM R/I or multiple tyrosine kinase inhibitor (Multi-TKI): IM, D and/or NI R/I.
- BP-CML Total (Part 2): All participants who received bosutinib 500 mg orally once daily in blast phase (BP) CML who were IM R/I or Multi-TKI: IM, D and/or NI R/I.
- Bosutinib 500 mg, Ph+ ALL (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with Ph+ ALL
Period: Period 1: Part 1 (Dose Escalation)
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1) | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Started | 3 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Continued in to Part 2 | 3 | 3 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2: Part 2 (Efficacy)
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1) | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Started | 0 | 0 | 0 | 195 (17 participants from Part 1 (Bosutinib 400mg, 500mg, 600mg cohort) continued in Part 2 of the study.) | 89 | 5 | 38 | 50 | 26 | 79 (1 participant from Part 1 (Bosutinib 600mg cohort) continued in Part 2 of the study.) | 64 | 24
Completed | 0 | 0 | 0 | 60 | 39 | 3 | 16 | 21 | 12 | 30 | 15 | 1
Not Completed | 0 | 0 | 0 | 135 | 50 | 2 | 22 | 29 | 14 | 49 | 49 | 23
Not completed — Discontinuation of study by sponsor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 9 | 8 | 1 | 3 | 3 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 12 | 4 | 0 | 4 | 0 | 1 | 4 | 4 | 0
Not completed — Other | 0 | 0 | 0 | 15 | 4 | 0 | 1 | 5 | 4 | 4 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 37 | 7 | 1 | 10 | 12 | 3 | 30 | 44 | 22
Not completed — Extension study | 0 | 0 | 0 | 61 | 27 | 0 | 4 | 9 | 5 | 9 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All-treated population - included all enrolled participants who received at least one dose of bosutinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2) | Total
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 79 | 64 | 24 | 570
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 73 | 22 | 1 | 5 | 7 | 10 | 26 | 29 | 6 | 179
  Between 45 and 64 years | 86 | 40 | 3 | 23 | 29 | 14 | 45 | 25 | 7 | 272
  >=65 years | 36 | 27 | 1 | 10 | 14 | 2 | 8 | 10 | 11 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 53 | 3 | 20 | 31 | 12 | 35 | 22 | 12 | 270
  Male | 113 | 36 | 2 | 18 | 19 | 14 | 44 | 42 | 12 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity, any clinically-significant grade 2 non-hematologic toxicity that requires 14 days to resolve (to grade 1).
Time Frame: Part 1 Baseline up to Day 28
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Bosutinib 400 mg (Part 1): Single oral dose of bosutinib 400 mg on Day 1 and then bosutinib 400 mg orally once daily continuously from Day 3 up to Week 4. All participants who completed treatment in Part 1 were continued in CP2L-CML Part 2 of the study.
- Bosutinib 600 mg (Part 1): Single oral dose of bosutinib 600 mg on Day 1 and then bosutinib 600 mg orally once daily continuously from Day 3 up to Week 4. All participants who completed treatment in Part 1 were continued in CP2L-CML Part 2 of the study. Eleven participants who completed treatment in Part 1 were continued in CP2L-CML Part 2 of the study and 1 participant was continued in AP-CML Part 2 of the study.
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
participants | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced DLT. DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity, any clinically-significant grade 2 non-hematologic toxicity that requires 14 days to resolve (to grade 1).
  NA = not estimable.
Time Frame: Part 1 Baseline up to Day 28
Population: Safety population included all participants who received at least 1 dose of study medication
Measure: Number; unit: mg
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
mg | NA — MTD was not achieved since no more than 1 DLT was observed in any cohort. At the 600mg dose level, 1 DLT and several treatment related grade 2 toxicities were observed, thus, Bosutinib 500 mg was selected as the recommended dose for part 2. | NA — MTD was not achieved since no more than 1 DLT was observed in any cohort. At the 600mg dose level, 1 DLT and several treatment related grade 2 toxicities were observed, thus, Bosutinib 500 mg was selected as the recommended dose for part 2. | NA — MTD was not achieved since no more than 1 DLT was observed in any cohort. At the 600mg dose level, 1 DLT and several treatment related grade 2 toxicities were observed, thus, Bosutinib 500 mg was selected as the recommended dose for part 2.

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) - Part 1
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: Evaluable population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
nanogram per milliliter (ng/mL) | 89.3 (50.0) | 101.0 (35.6) | 120.0 (40.2)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) - Part 1
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: Evaluable population included all enrolled participants who received at least one dose of study medication and had an adequate baseline efficacy assessment.
Measure: Median (Full Range); unit: hours (hrs)
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
hours (hrs) | 4.00 [3.33 to 48.08] | 6.00 [6.00 to 6.00] | 4.00 [2.17 to 49.33]

5. Primary Outcome: Plasma Decay Half-Life (t1/2) - Part 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
  NA = not estimable.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: Evaluable population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline efficacy assessment. 'N' (number of participants analyzed) signifies number of participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 2 | 3 | 8
hrs | 22.91 (3.39) | 22.46 (1.73) | 22.24 (5.03)

6. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC(0-48)] - Part 1
Description: AUC(0-48)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-48).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
ng*hr/mL | 1850 (710) | 2060 (483) | 2340 (1140)

7. Primary Outcome: Area Under the Concentration-Time Curve (AUC) - Part 1
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
  NA = not estimable.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 2 | 3 | 8
ng*hr/mL | 2530 (1160) | 2760 (687) | 2420 (457)

8. Primary Outcome: Apparent Oral Clearance (CL/F) - Part 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
  NA = not estimable.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 2 | 3 | 8
liter per hour (L/hr) | 177 (81.3) | 189 (47.5) | 258 (61.2)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F) - Part 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24, 48 hours post-dose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 8
liter | 6050 (3550) | 6080 (1230) | 8540 (3820)

10. Primary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss) - Part 1
Description: Maximum plasma concentration over 24 hours at steady state (ss), on Day 15.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 10
ng/mL | 146 (20.0) | 200 (11.9) | 208 (73.3)

11. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax,ss) - Part 1
Description: Time to reach maximum observed plasma concentration over 24 hours at steady state (ss), on Day 15.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 15
Population: as for outcome 3
Measure: Median (Full Range); unit: hrs
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
hrs | 4.05 [3.08 to 6.08] | 6.05 [4.00 to 8.00] | 6.00 [2.83 to 11.08]

12. Primary Outcome: Plasma Decay Half-Life at Steady State (t1/2,ss) - Part 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Plasma decay half-life over 24 hours at steady state (ss), on Day 15 was calculated.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 7
hrs | 45.96 (32.30) | 21.71 (4.64) | 25.87 (24.85)

13. Primary Outcome: Area Under the Concentration-Time Curve at Steady State (AUCss) - Part 1
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. AUC over 24 hours at steady state (ss), on Day 15 was calculated.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 9
ng*hr/mL | 2720 (442) | 3650 (425) | 3630 (1270)

14. Primary Outcome: Apparent Oral Clearance at Steady State (CL/F,ss) - Part 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Apparent oral clearence over 24 hours at steady state (ss), on Day 15 was calculated.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 9
L/hr | 150 (23.2) | 138 (16.6) | 185 (66.2)

15. Primary Outcome: Accumulation Ratio (R)
Description: R=accumulation ratio (AUCss on Day 15/AUC0-24 on Day 1)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 1 and Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 9
ratio | 3.1 (1.4) | 2.8 (0.8) | 2.5 (0.9)

16. Primary Outcome: Percentage of Participants With MCyR at Week 24 in Chronic Phase Second-line Imatinib Resistant CML Population - Part 2
Description: CyR is based on the prevalence of Ph+ cells. Major cytogenetic response was categorized as either CCyR or partial CyR (PCyR). CCyR was achieved when there was 0 percent (%) Ph+ cells from at least 20 metaphases from conventional bone marrow cytogenetics or less than (<) 1% positive cells from at least 200 cells analyzed from fluorescent in situ hybridization (FISH). PCyR was achieved when 1 to 35% Ph+ cells were present.
Time Frame: Week 24
Population: Cytogenetic evaluable population included all enrolled participants who received at least one dose of study medication and had an adequate baseline cytogenetic assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2)
Number analyzed (Participants) | 182
percentage of participants | 35.7 [28.8 to 43.1]

17. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) - Part 1
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells. Major cytogenetic response was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR was achieved when there was 0% Ph+ cells from at least 20 metaphases from conventional bone marrow cytogenetics or <1% positive cells from at least 200 cells analyzed from FISH. PCyR was achieved when 1 to 35% Ph+ cells were present.
Time Frame: Weeks 12, 24, 36, 48 and the end of active treatment phase of Part 1 (Week 52)
Population: Cytogenetic evaluable population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline cytogenetic assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 3 | 3 | 12
percentage of participants | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 50.0 [21.1 to 78.9]

18. Secondary Outcome: Phosphorylation Inhibition of Breakpoint Cluster Region-Abelson Kinase (Bcr-Abl) - Part 1
Description: bcr-Abl is a protein resulting from the transcription of the Philadelphia chromosome following 9:22 chromosomal translocation, and phosphorylation inhibition of which correlates with inhibition of tumor cell growth.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 48 and the end of the active treatment phase of Part 1 (Week 52)
Population: Data was not summarized since inadequate data included the issue that molecular transcript analyses could not be performed, because of potential sample quality issues due to time required to transport the specimens from the few investigational sites to the central laboratory.
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Phosphorylation Inhibition of Crk Like (CrkL) Protein at Baseline - Part 1
Description: CrkL is a protein, phosphorylation of which has been shown to correlate with CML cell growth; and conversely inhibition of their phosphorylation correlates with inhibition of tumor cell growth. Phosphorylation of CrkL was monitored in whole blood cells, as well as in the cluster of differentiation 3 (CD3+) (T cell), CD19+ (B cell) and CD34+ (blast cell) compartments by using fluorescent activated cell sorter (FACS) flow cytometry.
Time Frame: 0 (pre-dose) on Day 1 (Baseline)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mol/100 cells
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 2 | 3 | 10
mol/100 cells | 457075 (559841.90) | 297967.33 (171643.30) | 397795.40 (552536.90)

20. Secondary Outcome: Percent Change From Baseline in Phosphorylation Inhibition of Crk Like Protein (CrkL) at Day 1, 8 and 15 - Part 1
Description: CrkL is a protein, phosphorylation of which has been shown to correlate with CML cell growth; and conversely inhibition of their phosphorylation correlates with inhibition of tumor cell growth. Phosphorylation of CrkL was monitored in whole blood cells, as well as in the CD3+ (T cell), CD19+ (B cell) and CD34+ (blast cell) compartments by using FACS flow cytometry.
  NA = not estimable.
Time Frame: 6 hours post-dose on Day 1, 0 (pre-dose), 6 hours post-dose on Day 8, 15
Population: Evaluable population included all enrolled participants who received at least 1 dose of study medication and had an adequate baseline efficacy assessment. 'N' signifies number of participants who were evaluable for this measure. n=number of participants evaluable for this measure at specified time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Bosutinib 400 mg (Part 1) | Bosutinib 500 mg (Part 1) | Bosutinib 600 mg (Part 1)
Number analyzed (Participants) | 1 | 3 | 9
percent change
  Day 1: post-dose (n=1, 1, 9) | -34.66 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 287.52 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 97.79 (283.61)
  Day 8: pre-dose (n=1, 1, 9) | 562.48 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 170.83 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 3.88 (128.97)
  Day 8: post-dose (n=1, 1, 9) | 528.62 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 429.79 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 143.57 (289.18)
  Day 15: pre-dose (n=1, 2, 7) | 177.87 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -44.64 (8.56) | 119.23 (170.91)
  Day 15: post-dose (n=1, 3, 7) | -49.85 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | -21.13 (57.91) | 138.45 (278.24)

21. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) in Chronic Phase Second-line and Chronic Phase Third-line CML Population - Part 2
Description: CyR is based on the prevalence of Ph+ cells. MCyR was categorized as either CCyR or PCyR. CCyR was achieved when there was 0% Ph+ cells from at least 20 metaphases from conventional bone marrow cytogenetics or <1% positive cells from at least 200 cells analyzed from FISH. PCyR was achieved when 1 to 35% Ph+ cells were present.
Time Frame: Week 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter up to Year 4 (CP3L) or Year 5 (CP2L)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-R (Part 2)
Number analyzed (Participants) | 80 | 5 | 36 | 45 | 26 | 182
percentage of participants | 61.3 [49.7 to 71.9] | 40.0 [5.3 to 85.3] | 38.9 [23.1 to 56.5] | 42.2 [27.7 to 57.9] | 38.5 [20.2 to 59.4] | 58.8 [51.3 to 66.0]

22. Secondary Outcome: Kaplan-Meier Estimate of Retaining an Attained/Maintained Major Cytogenetic Response (MCyR) at Year 5 in Chronic Phase Second-line CML - Part 2
Description: MCyR was categorized as either CCyR or PCyR. CCyR was achieved when there was 0% Ph+ cells from at least 20 metaphases from conventional bone marrow cytogenetics or <1% positive cells from at least 200 cells analyzed from FISH. PCyR was achieved when 1 to 35% Ph+ cells were present. The Kaplan-Meier probability of retaining an attained/maintained MCyR at Year 5 is reported. Median durations were not reached as of the minimum follow-up. Duration of response in weeks =(date of confirmed loss of first attained response or last valid cytogenetic assessment for those censored - date of first attained response)/7.
Time Frame: From first MCyR to loss of MCyR or censoring, assessed every 12 weeks up to 2 years and then every 24 weeks thereafter up to Year 5
Population: Subgroup of participants from evaluable population who had MCyR.
Measure: Number (95% Confidence Interval); unit: % probability of retaining MCyR
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2)
Number analyzed (Participants) | 107 | 49
% probability of retaining MCyR | 67.2 [56.8 to 75.6] | 79.8 [63.1 to 89.5]

23. Secondary Outcome: Time to Achieve Major Cytogenetic Response (MCyR) in Chronic Phase Second-line CML for Responders Only - Part 2
Description: MCyR was categorized as either CCyR or PCyR. CCyR was achieved when there was 0% Ph+ cells from at least 20 metaphases from conventional bone marrow cytogenetics or <1% positive cells from at least 200 cells analyzed from FISH. PCyR was achieved when 1 to 35% Ph+ cells were present. Time to MCyR was the interval from the date of first dose of study medication until the first date of achieving a given response.
  Time to response in weeks equals (=) (event date minus (-) first dose date plus (+) 1)divided (/)7, where the event date is the non-missing date of the first attained response for responders only.
Time Frame: Week 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter up to Year 5
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2)
Number analyzed (Participants) | 107 | 49
weeks | 12.3 [12.1 to 24.0] | 12.1 [12.0 to 12.3]

24. Secondary Outcome: Kaplan-Meier Estimate of Maintaining Complete Hematologic Response (CHR) at Year 4 (CP3L and ADV) or Year 5 (CP2L) - Part 2
Description: Hematologic response: if participants met all of the following criteria of CHR: White Blood Cells equal to or less than (≤) institutional upper limit of normal, no peripheral blood blasts or promyelocytes, myelocytes+metamyelocytes <5% in blood, absolute neutrophil count greater than or equal to (≥) 1.0×10^9 per liter (/L) , platelets ≥100×10^9/L & <450×10^9/L, <20% basophils in blood & no extramedually involvement (including hepato- or splenomegaly), ≤5% BM blasts (ADV only & applicable to CP if BM aspirate was performed). The duration of CHR was defined as the interval from the first date of response until the first date of confirmed loss of response. Duration of response in weeks =(date of confirmed loss of attained response or last valid hematologic assessment for those censored - date of first confirmed response)/7. The Kaplan-Meier estimate of maintaining CHR at the end of minimum follow-up is presented (CP2L: Year 5; CP3L & ADV: Year 4). NA = not estimable.
  NA = not estimable.
Time Frame: From date of first confirmed CHR to loss of CHR or censoring, assessed at Day 1 and 7 of Week 1, Day 7 of Week 2, 3, 4, 8, 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter up to Year 4 (CP3L and ADV) or Year 5 (CP2L)
Population: Subgroup of participants from evaluable population who had confirmed CHR.
Measure: Number (95% Confidence Interval); unit: % estimate of maintaining response
Groups:
- Bosutinib 500 mg, AP-CML IM R/I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with AP IM R/I CML; who had no prior proto-oncogene tyrosine-protein kinase Src, Abl, or Src-Abl inhibitor exposure other than IM.
- Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with AP Multi-TKI: IM, D and/or NI R/I CML.
- Bosutinib 500 mg, BP-CML IM R/I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with BP IM R/I CML ; who had no prior proto-oncogene tyrosine-protein kinase Src, Abl, or Src-Abl inhibitor exposure other than IM.
- Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2): Bosutinib 500 mg was administered orally once-daily in participants with BP Multi-TKI: IM, D and/or NI R/I CML.
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 169 | 76 | 4 | 26 | 37 | 19 | 17 | 7 | 9 | 1 | 2
% estimate of maintaining response | 61.5 [52.9 to 69.1] | 78.2 [64.4 to 87.1] | 50.0 [5.8 to 84.5] | 56.5 [30.9 to 75.8] | 69.9 [49.7 to 83.3] | 61.9 [33.6 to 81.0] | 47.1 [20.7 to 69.7] | 64.3 [15.1 to 90.2] | NA [NA to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | NA [NA to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | 100 [NA to 100] — Lower limit of the 95% CI was NA due to insufficient patients and/or follow-up.

25. Secondary Outcome: Duration of Complete Hematologic Response (CHR) - Part 2
Description: Hematologic response: if participants met all of the following criteria of CHR: White Blood Cells equal to or less than (≤) institutional upper limit of normal, no peripheral blood blasts or promyelocytes, myelocytes+metamyelocytes less than (<)5% in blood, absolute neutrophil count greater than or equal to (≥) 1.0×10^9 per liter (/L) , platelets <450×10^9/L, platelets ≥100×10^9/L, <20% basophils in blood and no extramedually involvement (including hepato- or splenomegaly), ≤5% BM blasts (required for ADV only and applicable to CP if BM aspirate was performed). The duration of CHR was defined as the interval from the first date of response until the first date of confirmed loss of response. Duration of response in weeks =(date of confirmed loss of attained response or last valid hematologic assessment for those censored - date of first confirmed response)/7.
  NA = not estimable.
Time Frame: as for outcome 24
Population: Subgroup of participants from evaluable population who had confirmed CHR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 169 | 76 | 4 | 26 | 37 | 19 | 17 | 7 | 9 | 1 | 2
weeks | NA [297.7 to NA] — KM estimate at Year 5 was NA due to insufficient patients and/or follow-up. The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 350.4 [350.4 to NA] — The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [9.6 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [38.3 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 295.6 [289.0 to NA] — The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [56.0 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 138.0 [24.0 to NA] — The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [102.0 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 28.6 [20.1 to NA] — The upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 40.0 [NA to NA] — 95% CIs were NA due to insufficient patients and/or follow-up. | NA [NA to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up.

26. Secondary Outcome: Time to Achieve Complete Hematologic Response (CHR) for Responders Only - Part 2
Description: The time to CHR was measured from the date of first dosing to the first date of response. Time to response in weeks = (event date - first dose date plus 1)/7, where the event date is the non-missing date of the first attained response for responders only.
Time Frame: Day 1 and 7 of Week 1, Day 7 of Week 2, 3, 4, 8, 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter up to Year 4 (CP3L and ADV) or Year 5 (CP2L)
Population: Hematologic evaluable population included all enrolled participants who received at least one dose of study medication and had an adequate baseline hematologic assessment - responders only.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 169 | 76 | 4 | 26 | 37 | 19 | 17 | 7 | 9 | 1 | 2
weeks | 2.0 [1.1 to 2.1] | 1.3 [1.1 to 2.1] | 1.6 [1.1 to 2.1] | 1.2 [1.1 to 3.0] | 1.3 [1.1 to 2.3] | 2.4 [1.1 to 3.3] | 12.1 [8.1 to 24.0] | 12.1 [4.3 to 72.0] | 8.0 [4.0 to 13.0] | 12.1 [NA to NA] — 95% CIs were NA due to insufficient patients and/or follow-up. | 10.0 [4.0 to 13.0]

27. Secondary Outcome: Cumulative Incidence of Progression/Death - Part 2
Description: The cumulative incidence of on-treatment progression or death adjusting for the competing risk of treatment discontinuation without the event. Disease progression was determined by the investigator as the reason for treatment discontinuation and death was due to any cause within 30 days of last dose. Duration in months = (date of PD/death or last valid cytogenetic/hematologic assessment if censored - first dose date)/30.4. 95% confidence intervals were calculated using Gray's method.
  NA = not estimable. One year = 12 months.
Time Frame: Years 1, 2, 3, 4, and 5 (CP2L only)
Population: All-treated population included all enrolled participants who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
percentage of participants
  Year 1 | 10.8 [7.2 to 16.1] | 4.5 [1.7 to 11.7] | 20.0 [3.5 to 100.0] | 23.7 [13.4 to 41.9] | 12.0 [5.7 to 25.4] | 23.1 [11.4 to 46.6] | 28.6 [18.4 to 44.5] | 20.0 [9.8 to 40.9] | 47.2 [33.4 to 66.7] | 71.4 [56.5 to 90.3] | 58.3 [41.6 to 81.8]
  Year 2 | 19.0 [14.2 to 25.4] | 6.7 [3.1 to 14.6] | 40.0 [13.7 to 100.0] | 23.7 [13.4 to 41.9] | 14.0 [7.0 to 27.8] | 30.8 [17.3 to 54.8] | 42.9 [31.0 to 59.2] | 23.3 [12.2 to 44.6] | 50.0 [36.1 to 69.3] | 71.4 [56.5 to 90.3] | 58.3 [41.6 to 81.8]
  Year 3 | 22.1 [16.9 to 28.7] | 9.0 [4.6 to 17.4] | 40.0 [13.7 to 100.0] | 23.7 [13.4 to 41.9] | 16.0 [8.5 to 30.2] | 34.6 [20.4 to 58.7] | 44.9 [32.9 to 61.2] | 26.7 [14.7 to 48.3] | 50.0 [36.1 to 69.3] | 75.0 [60.6 to 92.9] | 58.3 [41.6 to 81.8]
  Year 4 | 22.6 [17.4 to 29.3] | 9.0 [4.6 to 17.4] | 40.0 [13.7 to 100.0] | 23.7 [13.4 to 41.9] | 16.0 [8.5 to 30.2] | 34.6 [20.4 to 58.7] | 44.9 [32.9 to 61.2] | 26.7 [14.7 to 48.3] | 50.0 [36.1 to 69.3] | 75.0 [60.6 to 92.9] | 58.3 [41.6 to 81.8]
  Year 5 | 23.1 [17.9 to 29.8] | 10.1 [5.4 to 18.8] | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4.

28. Secondary Outcome: Progression Free Survival (PFS) - Part 2
Description: PFS was based on Kaplan-Meier method. Disease progression was determined by the investigator as the reason for treatment discontinuation and death was due to any cause within 30 days of last dose. Duration in months = (date of PD/death or last valid cytogenetic/hematologic assessment if censored - first dose date)/30.4.
  NA = not estimable. One year = 12 months
Time Frame: Years 1, 2, 3, 4, and 5 (CP2L only)
Population: All-treated population included all enrolled participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
Months | NA [NA to NA] — KM estimate at Year 5 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | 81.5 [81.5 to NA] — Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [0.9 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [11.1 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [68.5 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | NA [14.1 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 20.4 [11.8 to NA] — Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 35.4 [14.6 to NA] — Upper limit of 95% CI was NA due to insufficient patients and/or follow-up. | 7.9 [4.0 to 10.1] | 1.8 [0.9 to 5.5] | 1.5 [0.7 to 3.8]

29. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) - Part 2
Description: OS was based on Kaplan-Meier method. Survival was defined as the time period from the date of first dose of bosutinib to the date of death or date of last contact for those censored.
  NA = not estimable. One year = 12 months.
Time Frame: Years 1, 2, 3, 4, and 5 (CP2L only)
Population: All-treated population included all enrolled participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
percentage of participants
  Year 1 | 96.3 [92.5 to 98.2] | 98.9 [92.1 to 99.8] | 100 [100 to 100] | 85.8 [69.2 to 93.8] | 91.8 [79.7 to 96.6] | 96.2 [75.7 to 99.4] | 81.3 [67.2 to 89.8] | 72.9 [53.0 to 85.4] | 44.3 [27.4 to 59.9] | 39.3 [21.7 to 56.5] | 16.7 [5.2 to 33.7]
  Year 2 | 88.2 [82.7 to 92.1] | 97.7 [91.0 to 99.4] | 80.0 [20.4 to 96.9] | 79.7 [62.0 to 89.8] | 83.3 [69.3 to 91.3] | 92.3 [72.6 to 98.0] | 72.7 [57.6 to 83.1] | 59.0 [39.2 to 74.3] | 41.3 [24.9 to 57.0] | 25.0 [11.1 to 41.8] | 8.3 [1.4 to 23.3]
  Year 3 | 84.1 [77.8 to 88.7] | 93.0 [83.9 to 97.1] | 80.0 [20.4 to 96.9] | 66.1 [44.5 to 80.9] | 83.3 [69.3 to 91.3] | 86.5 [62.9 to 95.6] | 70.1 [54.7 to 81.1] | 45.1 [25.4 to 63.0] | 41.3 [24.9 to 57.0] | 16.7 [5.6 to 32.9] | 8.3 [1.4 to 23.3]
  Year 4 | 81.5 [74.7 to 86.6] | 93.0 [83.9 to 97.1] | 80.0 [20.4 to 96.9] | 66.1 [44.5 to 80.9] | 79.3 [63.1 to 89.0] | 86.5 [62.9 to 95.6] | 65.7 [48.6 to 78.3] | 45.1 [25.4 to 63.0] | 20.7 [2.0 to 53.2] | 16.7 [5.6 to 32.9] | 8.3 [1.4 to 23.3]
  Year 5 | 80.6 [73.6 to 85.9] | 88.4 [76.6 to 94.5] | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4. | NA [NA to NA] — In Part 2 subjects in CP3L and ADV treatment groups were only evaluated up to Year 4.

30. Secondary Outcome: Overall Survival (OS) - Part 2
Description: as for outcome 29
Time Frame: Years 1, 2, 3, 4, and 5 (CP2L only)
Population: All-treated population included all enrolled participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
Months | NA [NA to NA] — KM estimate at Year 5 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | 81.5 [81.5 to NA] — The upper 95% CI was NA due to insufficient patients and/or follow-up. | NA [21.0 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper 95% CI was NA due to insufficient patients and/or follow-up. | NA [34.4 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper 95% CI was NA due to insufficient patients and/or follow-up. | NA [68.5 to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. The upper 95% CI was NA due to insufficient patients and/or follow-up. | NA [NA to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | NA [NA to NA] — KM estimate at Year 4 was NA due to insufficient patients and/or follow-up. 95% CIs were NA due to insufficient patients and/or follow-up. | 33.4 [14.6 to NA] — The upper 95% CI was NA due to insufficient patients and/or follow-up. | 11.2 [9.4 to NA] — The upper 95% CI was NA due to insufficient patients and/or follow-up. | 8.9 [4.1 to 17.4] | 3.6 [1.3 to 7.6]

31. Secondary Outcome: Percentage of Participants With Confirmed Complete Hematologic Response (CHR) - Part 2
Description: Hematologic response: if participants met all of the following criteria of CHR: White Blood Cells ≤ institutional upper limit of normal, no peripheral blood blasts or promyelocytes, myelocytes+metamyelocytes <5% in blood, absolute neutrophil count ≥ 1.0×10^9/L , platelets <450×10^9/L, platelets ≥100×10^9/L, <20% basophils in blood and no extramedually involvement (including hepato- or splenomegaly), ≤5% BM blasts (required for ADV only and applicable to CP if BM aspirate was performed).
Time Frame: as for outcome 26
Population: Hematologic evaluable population included all enrolled participants who received at least one dose of study medication and had an adequate baseline hematologic assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 194 | 89 | 5 | 38 | 49 | 25 | 43 | 29 | 34 | 26 | 22
percentage of participants | 87.1 [81.6 to 91.5] | 85.4 [76.3 to 92.0] | 80.0 [28.4 to 99.5] | 68.4 [51.3 to 82.5] | 75.5 [61.1 to 86.7] | 76.0 [54.9 to 90.6] | 39.5 [25.0 to 55.6] | 24.1 [10.3 to 43.5] | 26.5 [12.9 to 44.4] | 3.8 [0.1 to 19.6] | 9.1 [1.1 to 29.2]

32. Secondary Outcome: Percentage of Participants With Overall Hematologic Response (OHR) by Week 48 in Advanced Leukemia Population - Part 2
Description: OHR included CHR, no evidence of leukemia (≤5% bone marrow blasts, no peripheral blood blasts or promyelocytes, <5% myelocytes + metamyelocytes in blood, white blood cells ≤ institutional upper limit of normal, 450x10^9/L > platelets > 20x10^9/L, absolute neutrophil count ≥0.5x10^9/L, <20% basophils in blood, no extramedullary involvement [including liver or spleen]), minor hematologic response (acute lymphoblastic leukemia [ALL] patients only, defined as <15% blasts in marrow & blood, <30% blasts + promyelocytes in marrow & blood, <20% basophils in peripheral blood & no extramedullary disease other than spleen & liver) or return to chronic phase (AP/BP participants, defined as <15% blasts in both peripheral blood &bone marrow, <30% blasts + promyelocytes in both peripheral blood & bone marrow, <20% basophils in both peripheral blood & bone marrow, no extramedullary Involvement other than liver or spleen). Participants had to meet at least 1 criterion.
Time Frame: Day 1 and 7 of Week 1, Day 7 of Week 2, 3, 4, 8, 12, thereafter assessed every 12 weeks up to 1 year
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 43 | 29 | 34 | 26 | 22
percentage of participants | 67.4 [51.5 to 80.9] | 41.4 [23.5 to 61.1] | 38.2 [22.2 to 56.4] | 15.4 [4.4 to 34.9] | 9.1 [1.1 to 29.2]

33. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to follow up visit (30 days after last dose of study treatment)
Population: Safety population included all participants who receive at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
percentage of participants
  AEs | 99.5 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 97.2 | 100.0 | 95.8
  SAEs | 41.5 | 38.2 | 20.0 | 39.5 | 38.0 | 19.2 | 49.0 | 63.3 | 55.6 | 60.7 | 70.8

34. Secondary Outcome: Duration of Potentially Clinically Important (PCI) Adverse Events (AEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. The event did not necessarily have a causal relationship with the treatment. PCI AEs included anemia, alanine aminotranferase (ALT), aspartate aminotransferase (AST), cardiac, diarrhea, edema, effusion, gastrointestinal, hemorrhage, hypersensitivity, hypertension, infection, liver, myelosuppression, nausea, neutropenia, rash, renal, thrombocytopenia, vomiting, and vascular events. Duration of AE was calculated as (stop date minus start date) plus 1 for non-missing and non-partial dates.
  NA = not estimable.
Time Frame: Baseline up to follow-up visit (30 days after last dose of study treatment)
Population: Safety population included all participants who receive at least one dose of study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 79 | 64 | 24
days
  Anaemia | 14.0 [1 to 1373] | 36.0 [2 to 688] | 38.0 [38 to 38] | 19.0 [1 to 284] | 13.0 [6 to 271] | 61.0 [6 to 335] | 12.5 [1 to 502] | 4.0 [1 to 52] | 7.0 [1 to 20]
  ALT | 29.0 [1 to 775] | 15.0 [1 to 344] | NA [NA to NA] — No events therefore duration not available. | 21.5 [7 to 236] | 8.0 [5 to 87] | 21.0 [4 to 42] | 21.5 [7 to 252] | 7.5 [1 to 41] | 3.0 [1 to 5]
  AST | 29.0 [1 to 803] | 13.5 [1 to 330] | NA [NA to NA] — No events therefore duration not available. | 18.0 [14 to 22] | 8.5 [8 to 22] | 15.0 [8 to 21] | 14.0 [1 to 188] | 2.0 [2 to 2] | 5.0 [5 to 5]
  Diarrhoea | 1.0 [1 to 2174] | 2.0 [1 to 1121] | 2.0 [1 to 59] | 2.0 [1 to 189] | 2.0 [1 to 413] | 1.0 [1 to 289] | 2.0 [1 to 910] | 2.0 [1 to 211] | 3.0 [1 to 500]
  Effusion | 18.5 [1 to 1428] | 29.0 [5 to 657] | 79.5 [14 to 421] | 20.0 [7 to 842] | 28.0 [1 to 907] | 20.0 [5 to 258] | 21.0 [4 to 1536] | 58.0 [11 to 101] | 5.0 [4 to 25]
  Infection | 10.0 [1 to 1026] | 9.5 [1 to 546] | 11.5 [1 to 46] | 8.0 [1 to 85] | 9.0 [2 to 366] | 8.0 [1 to 183] | 9.0 [1 to 281] | 9.5 [1 to 78] | 9.0 [1 to 39]
  Nausea | 2.0 [1 to 972] | 4.0 [1 to 446] | 4.0 [1 to 7] | 2.0 [1 to 168] | 14.0 [1 to 713] | 2.0 [1 to 42] | 6.0 [1 to 247] | 6.5 [1 to 274] | 9.0 [1 to 31]
  Neutropenia | 23.0 [1 to 506] | 15.0 [1 to 337] | 23.0 [13 to 70] | 14.5 [4 to 81] | 21.0 [3 to 504] | 26.0 [7 to 92] | 8.0 [1 to 252] | 5.0 [1 to 52] | 6.5 [5 to 8]
  Oedema | 29.0 [1 to 1416] | 81.5 [1 to 1807] | 4.0 [1 to 52] | 1.0 [1 to 455] | 12.5 [2 to 774] | 28.0 [3 to 316] | 88.5 [2 to 670] | 11.0 [1 to 214] | 5.0 [1 to 8]
  Rash | 15.0 [1 to 1622] | 13.0 [1 to 965] | 17.0 [7 to 52] | 12.0 [1 to 348] | 19.0 [1 to 1612] | 12.5 [1 to 150] | 13.0 [1 to 428] | 7.5 [1 to 218] | 12.0 [1 to 33]
  Renal events | 27.0 [1 to 831] | 190.0 [7 to 903] | 1167.0 [1167 to 1167] | 162.0 [21 to 299] | 11.0 [1 to 203] | 56.5 [29 to 84] | 26.0 [3 to 1403] | 9.0 [1 to 27] | 12.0 [12 to 12]
  Thrombocytopenia | 22.0 [1 to 1762] | 15.0 [1 to 1541] | 38.5 [14 to 120] | 15.0 [1 to 336] | 15.0 [2 to 420] | 21.5 [6 to 350] | 11.5 [1 to 889] | 5.0 [1 to 176] | 9.0 [3 to 43]
  Vomiting | 1.0 [1 to 165] | 1.0 [1 to 36] | NA [NA to NA] — No events therefore duration not available. | 1.0 [1 to 141] | 2.0 [1 to 59] | 7.0 [1 to 39] | 1.0 [1 to 128] | 1.0 [1 to 41] | 1.5 [1 to 9]
  Cardiac events | 11.0 [1 to 1428] | 6.0 [1 to 657] | NA [NA to NA] — No events therefore duration not available. | 7.5 [1 to 842] | 22.0 [1 to 907] | 1.0 [1 to 1] | 14.0 [1 to 1536] | 3.0 [1 to 19] | 1.5 [1 to 2]
  Vascular events | 3.5 [1 to 277] | 6.0 [1 to 59] | NA [NA to NA] — No events therefore duration not available. | 10.5 [3 to 18] | 1.5 [1 to 266] | 10.0 [10 to 10] | 2.0 [1 to 22] | 1.0 [1 to 14] | 1.0 [1 to 19]
  Hypertension | 16.0 [1 to 1343] | 1.0 [1 to 1659] | NA [NA to NA] — No events therefore duration not available. | 7.0 [7 to 7] | 1.0 [1 to 418] | NA [NA to NA] — No events therefore duration not available. | 5.0 [1 to 204] | NA [NA to NA] — No events therefore duration not available. | 2.0 [2 to 2]
  Gastrointestinal events | 1.0 [1 to 2174] | 2.0 [1 to 1121] | 2.0 [1 to 59] | 2.0 [1 to 189] | 2.0 [1 to 713] | 2.0 [1 to 289] | 2.0 [1 to 910] | 3.0 [1 to 274] | 4.0 [1 to 500]
  Haemorrhage | 10.0 [1 to 862] | 16.0 [1 to 131] | 23.0 [23 to 23] | 4.0 [1 to 11] | 27.5 [1 to 190] | 7.5 [1 to 58] | 6.0 [1 to 147] | 4.0 [1 to 28] | 3.5 [1 to 21]
  Hypersensitivity | 9.0 [6 to 38] | 8.0 [7 to 9] | NA [NA to NA] — No events therefore duration not available. | 7.0 [1 to 28] | 6.0 [1 to 15] | 5.0 [1 to 9] | 1.0 [1 to 1] | NA [NA to NA] — No events therefore duration not available. | NA [NA to NA] — No events therefore duration not available.
  Liver | 29.0 [1 to 803] | 16.0 [1 to 344] | 8.0 [8 to 8] | 25.5 [7 to 236] | 9.0 [5 to 136] | 21.0 [3 to 82] | 16.0 [1 to 252] | 8.0 [1 to 441] | 5.0 [1 to 9]
  Myelosuppression | 22.0 [1 to 1762] | 18.0 [1 to 1541] | 28.0 [13 to 120] | 15.0 [1 to 336] | 15.0 [2 to 504] | 27.0 [6 to 769] | 11.5 [1 to 889] | 5.0 [1 to 376] | 7.0 [1 to 43]

35. Secondary Outcome: Percentage of Participants With Change From Baseline in Laboratory Tests Results
Description: Laboratory assessments included urinalysis, complete blood count (CBC), prothrombin time/partial prothromboplastin time (PT/PPT), international normalized ratio (INR), blood chemistry and serum pregnancy test (β-HCG). Parameters of special interest included liver function tests and those related to myelosuppression. Potentially clinically important (PCI) laboratory values were defined as National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE v3.0) grade 3 or higher. Maximum CTCAE grade, and only participants who shifted to Grade 3/4 on-treatment, are reported.
Time Frame: Week 1, 2, 3, 4, 8, 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter
Population: Safety population included all participants who receive at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 79 | 64 | 24
Percentage of Participants
  Hemoglobin: shift from Normal to Grade 3 | 0.5 | 1.1 | 0.0 | 0.0 | 0.0 | 3.8 | 5.1 | 1.6 | 0.0
  Hemoglobin: shift from Normal to Grade 4 | 1.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin: shift from Grade 1 to Grade 3 | 3.6 | 10.1 | 0.0 | 2.6 | 0.0 | 0.0 | 7.6 | 6.3 | 8.3
  Hemoglobin: shift from Grade 1 to Grade 4 | 1.5 | 0.0 | 0.0 | 0.0 | 4.0 | 0.0 | 1.3 | 3.1 | 0.0
  Hemoglobin: shift from Grade 2 to Grade 3 | 3.1 | 6.7 | 0.0 | 7.9 | 0.0 | 0.0 | 10.1 | 15.6 | 16.7
  Hemoglobin: shift from Grade 2 to Grade 4 | 2.1 | 1.1 | 0.0 | 0.0 | 4.0 | 0.0 | 2.5 | 4.7 | 4.2
  Hemoglobin: shift from Grade 3 to Grade 4 | 0.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 5.1 | 4.7 | 0.0
  Absolute neutrophils (ANC): Normal to Grade 3 | 7.2 | 9.0 | 0.0 | 5.3 | 4.0 | 11.5 | 10.1 | 3.1 | 0.0
  ANC: shift from Normal to Grade 4 | 2.1 | 3.4 | 20.0 | 7.9 | 4.0 | 3.8 | 2.5 | 3.1 | 0.0
  ANC: shift from Grade 1 to Grade 3 | 0.0 | 2.2 | 0.0 | 0.0 | 0.0 | 0.0 | 2.5 | 7.8 | 12.5
  ANC: shift from Grade 1 to Grade 4 | 0.5 | 0.0 | 0.0 | 2.6 | 2.0 | 0.0 | 1.3 | 20.3 | 4.2
  ANC: shift from Grade 2 to Grade 3 | 1.0 | 3.4 | 0.0 | 2.6 | 2.0 | 0.0 | 3.8 | 0.0 | 0.0
  ANC: shift from Grade 2 to Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.3 | 3.1 | 8.3
  ANC: shift from Grade 3 to Grade 4 | 0.0 | 1.1 | 0.0 | 0.0 | 2.0 | 0.0 | 0.0 | 4.7 | 8.3
  Platelet count: shift from Normal to Grade 3 | 13.3 | 13.5 | 0.0 | 15.8 | 12.0 | 7.7 | 11.4 | 4.7 | 4.2
  Platelet count: shift from Normal to Grade 4 | 3.6 | 7.9 | 0.0 | 0.0 | 8.0 | 15.4 | 7.6 | 1.6 | 0.0
  Platelet count: shift from Grade 1 to Grade 3 | 3.6 | 5.6 | 0.0 | 2.6 | 2.0 | 3.8 | 5.1 | 3.1 | 4.2
  Platelet count: shift from Grade 1 to Grade 4 | 1.5 | 1.1 | 0.0 | 2.6 | 4.0 | 0.0 | 6.3 | 6.3 | 0.0
  Platelet count: shift from Grade 2 to Grade 3 | 0.5 | 2.2 | 20.0 | 0.0 | 2.0 | 0.0 | 3.8 | 4.7 | 0.0
  Platelet count: shift from Grade 2 to Grade 4 | 0.5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.3 | 4.7 | 0.0
  Platelet count: shift from Grade 3 to Grade 4 | 1.0 | 0.0 | 0.0 | 0.0 | 2.0 | 0.0 | 5.1 | 10.9 | 29.2
  ALT: shift from Normal to Grade 3 | 8.7 | 12.4 | 0.0 | 0.0 | 10.0 | 15.4 | 5.1 | 1.6 | 0.0
  ALT: shift from Grade 1 to Grade 3 | 1.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.8 | 0.0 | 0.0
  AST: shift from Normal to Grade 3 | 4.1 | 7.9 | 0.0 | 0.0 | 0.0 | 7.7 | 2.5 | 1.6 | 0.0
  AST: shift from Normal to Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.8 | 0.0 | 0.0 | 0.0
  AST: shift from Grade 1 to Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 2.0 | 0.0 | 2.5 | 0.0 | 0.0
  ALP: shift from Normal to Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.3 | 0.0 | 0.0
  ALP: shift from Grade 1 to Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.6 | 0.0
  Total bilirubin: shift from Normal to Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 2.0 | 0.0 | 0.0 | 6.3 | 4.2
  ALT: shift from Normal to Grade 4 | 0.0 | 2.2 | 0.0 | 0.0 | 0.0 | 3.8 | 0.0 | 0.0 | 0.0
  Total bilirubin: shift from Grade 2 to Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 2.0 | 0.0 | 0.0 | 0.0 | 0.0

36. Secondary Outcome: Percentage of Participants With On-treatment PCI Change From Baseline in Electrocardiogram (ECG) Findings
Description: Criteria for PCI changes in ECG (12-lead) were defined as: no sinus rhythm; PR interval >=220 msec and increase of >=20 msec; QRS interval >=120 msec; QT interval corrected using the Fridericia formula (QTcF) and QT interval corrected using the Bazett formula (QTcB) >500 msec or increase of >60 msec; heart rate <=45 beats per minute (bpm) or >=120 bpm or decrease/increase of >=15 bpm.
Time Frame: Baseline, 0 (pre-dose), 2, 4, 6 hours on Day 1, 0 (pre-dose), 2, 4, 6, 20-23 hours on Day 21, and end of treatment visit
Population: Safety population included all participants who receive at least one dose of study medication. 'N' (Number of Participants Analyzed) signifies number of participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 37 | 50 | 26 | 78 | 62 | 23
Percentage of participants | 32.3 | 23.6 | 20.0 | 24.3 | 22.0 | 23.1 | 39.7 | 59.7 | 34.8

37. Secondary Outcome: Number of Participants With Change From Baseline in Findings of Chest X-ray
Description: Number of participants whose chest X-ray results changed (worsened or improved) from the Baseline.
Time Frame: Baseline, Week 8, and end of treatment
Population: Safety population included all participants who received at lease one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 79 | 64 | 24
participants
  Worsened From Baseline | 35 | 18 | 1 | 6 | 18 | 3 | 16 | 10 | 3
  Improved From Baseline | 15 | 7 | 0 | 4 | 1 | 3 | 6 | 11 | 1
  Total | 50 | 25 | 1 | 10 | 19 | 6 | 22 | 21 | 4

38. Secondary Outcome: Number of Participants Who Received Concomitant Medications for Management of Adverse Events (AEs)
Description: Number of participants taking any non-study medications which were administered from Study Day 1 to 30 days after last dose of study treatment as a management of an AE are reported.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 8, 12, then every 12 weeks thereafter until end of treatment, for a mean duration of 28 months
Population: Safety population included all participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 79 | 64 | 24
participants
  ALT | 7 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  AST | 5 | 3 | 0 | 2 | 3 | 4 | 2 | 0 | 0
  Anemia | 6 | 8 | 2 | 2 | 2 | 1 | 6 | 1 | 1
  Cardiac events | 13 | 4 | 0 | 2 | 6 | 0 | 7 | 2 | 1
  Gastrointestinal toxicity - Diarrhoea | 120 | 46 | 2 | 22 | 26 | 14 | 44 | 22 | 10
  Effusion | 11 | 5 | 1 | 3 | 9 | 1 | 9 | 2 | 0
  Haemorrhage | 12 | 3 | 0 | 1 | 0 | 1 | 4 | 6 | 3
  Hypertension | 15 | 4 | 0 | 2 | 4 | 1 | 7 | 2 | 2
  Hypersensitivity reactions | 5 | 2 | 0 | 4 | 2 | 2 | 1 | 1 | 0
  Infection | 92 | 39 | 4 | 11 | 18 | 10 | 37 | 30 | 7
  Hepatic events | 10 | 5 | 0 | 0 | 0 | 2 | 3 | 3 | 0
  Gastrointestinal toxicity - Nausea | 33 | 25 | 1 | 11 | 10 | 8 | 19 | 23 | 7
  Neutropenia | 2 | 5 | 1 | 5 | 1 | 1 | 6 | 5 | 2
  Rash | 44 | 37 | 2 | 8 | 16 | 3 | 20 | 9 | 2
  Oedema | 13 | 9 | 1 | 3 | 3 | 0 | 7 | 7 | 3
  Renal | 2 | 2 | 0 | 0 | 1 | 0 | 4 | 3 | 0
  Thrombocytopenia | 4 | 2 | 3 | 10 | 19 | 13 | 3 | 3 | 0
  Vascular events | 6 | 3 | 0 | 0 | 3 | 0 | 2 | 1 | 0
  Gastrointestinal toxicity - Vomiting | 25 | 9 | 0 | 5 | 7 | 4 | 17 | 14 | 4

39. Secondary Outcome: Number of Participants With Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG-PS)
Description: ECOG-PS measured on-therapy (time between first dose and last dose date with a 30-day lag) assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction;1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work;2=ambulatory (>50% of waking hrs), capable of all self care, unable to carry out any work activities;3=capable of only limited self care, confined to bed/chair >50% of waking hrs;4=completely disabled, cannot carry on any self care, totally confined to bed/chair;5=dead.
Time Frame: Baseline, Week 1, 2, 8, 12, thereafter assessed every 12 weeks up to 2 years then every 24 weeks thereafter
Population: Safety population included all participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | Bosutinib 500 mg, AP-CML IM R/I (Part 2) | Bosutinib 500 mg, AP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, BP-CML IM R/I (Part 2) | Bosutinib 500 mg, BP-CML Multi-TKI R/I (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 195 | 89 | 5 | 38 | 50 | 26 | 49 | 30 | 36 | 28 | 24
participants
  Baseline: Grade 0; maximum on-therapy: Grade 0 | 92 | 36 | 2 | 21 | 20 | 19 | 17 | 9 | 9 | 2 | 2
  Baseline: Grade 0; maximum on-therapy: Grade 1 | 50 | 25 | 0 | 5 | 8 | 5 | 11 | 5 | 47 | 2 | 4
  Baseline: Grade 0; maximum on-therapy: Grade 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
  Baseline: Grade 0; maximum on-therapy: Grade 3 | 4 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Baseline: Grade 0; maximum on-therapy: Grade 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Grade 1; maximum on-therapy: Grade 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 1
  Baseline: Grade 1; maximum on-therapy: Grade 1 | 32 | 13 | 2 | 7 | 13 | 2 | 14 | 7 | 7 | 5 | 3
  Baseline: Grade 1; maximum on-therapy: Grade 2 | 10 | 6 | 1 | 1 | 5 | 0 | 2 | 5 | 0 | 6 | 3
  Baseline: Grade 1; maximum on-therapy: Grade 3 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0
  Baseline: Grade 1; maximum on-therapy: Grade 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Baseline: Grade 2; maximum on-therapy: Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline: Grade 2; maximum on-therapy: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Baseline: Grade 2; maximum on-therapy: Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 4
  Baseline: Grade 2; maximum on-therapy: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
  Baseline: Grade 2; maximum on-therapy: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Baseline: Missing | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Grade 0; maximum on-therapy: Missing | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Baseline: Grade 1; maximum on-therapy: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

40. Secondary Outcome: Percentage of Participants With Change From Baseline in Physical Examinations and Vital Signs
Description: Percentage of participants with PCI physical examinations and vital signs is reported during therapy and at post therapy. Criteria for PCI change in vital signs: heart rate value of <40 beats per min and value >150 beats per min, systolic blood pressure (SBP) of <80 or >210 millimeter of mercury (mmHg), diastolic blood pressure (DBP) of <40 or >130 mmHg, temperature <32 or >40 degree centigrade, respiratory rate (Resp) of <10 or >50 breaths/min and criteria for PCI change in physical examination: >=10% increase or decrease of body weight in kilogram (kg).
Time Frame: Screening, Baseline, and end of treatment
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 188 | 81 | 5 | 35 | 46 | 25 | 75 | 56 | 20
percentage of participants
  SBP >210 mmHg | 1.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight increase 10% | 16.0 | 6.3 | 20.0 | 12.1 | 6.5 | 16.0 | 11.0 | 7.5 | 6.3
  Weight decrease 10% | 21.9 | 16.3 | 0 | 6.1 | 15.2 | 0 | 23.3 | 9.4 | 0
  SBP <80 mmHg | 0 | 0 | 0 | 0 | 0 | 4.0 | 0 | 0 | 0
  Temperature <32C | 0 | 0 | 0 | 0 | 0 | 4.0 | 0 | 0 | 0
  Pulse <40bpm | 0 | 1.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Resp >50 breaths/min | 0 | 0 | 0 | 0 | 0 | 5.0 | 0 | 0 | 0
  Resp <10 breaths/min | 0 | 0 | 0 | 0 | 2.4 | 0 | 0 | 0 | 0

41. Secondary Outcome: Percentage of Participants With Change From Baseline in Physical Examinations and Vital Signs and Number of Participants With PCI Values
Description: Percentage of participants with PCI physical examinations and vital signs is reported during therapy and at post therapy. Criteria for PCI change in vital signs: heart rate value of <40 beats per min and value >150 beats per min, SBP of <80 or >210 mmHg, DBP of <40 or >130 mmHg, temperature <32 or >40 degree centigrade, Resp of <10 or >50 breaths/min and criteria for PCI change in physical examination: >=10% increase or decrease of body weight in kg. No Ph+ ALL participants were analyzed post-therapy (N=0). Part 1 safety data were originally presented in 2011 and are included as cumulative data in the Part 2 final safety results.
Time Frame: Post-therapy
Population: Safety population included all participants who receive at least one dose of study medication. 'N' (number of participants analyzed) signifies number of participants who were evaluable for this measure. PLEASE NOTE: Results were not applicable for Arms in Part 1 since all participants in Part 1 entered Part 2 and continued the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Number analyzed (Participants) | 24 | 16 | 1 | 2 | 11 | 4 | 8 | 3 | 0
percentage of participants
  Pulse <40 bpm | 4.2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  SBP >210 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0 |
  Weight increase 10% | 4.2 | 0 | 0 | 0 | 0 | 0 | 0 | 33.3 |
  Weight decrease 10% | 12.5 | 6.7 | 0 | 0 | 9.1 | 0 | 16.7 | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs were assessed from informed consent through and including 30 days after last administration of study treatment or at the End of Treatment Visit, whichever comes last.
Description: An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. Part 1 safety data were originally presented in 2011 and are included as cumulative data in the Part 2 final safety results.
Arm/Group | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) | AP-CML Total (Part 2) | BP-CML Total (Part 2) | Bosutinib 500 mg, Ph+ ALL (Part 2)
Serious Adverse Events (participants affected / at risk) | 81/195 | 34/89 | 1/5 | 15/38 | 19/50 | 5/26 | 43/79 | 37/64 | 17/24
Other Adverse Events (participants affected / at risk) | 194/195 | 89/89 | 5/5 | 38/38 | 50/50 | 26/26 | 79/79 | 62/64 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) (N=195) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) (N=89) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) (N=5) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) (N=38) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) (N=50) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) (N=26) | AP-CML Total (Part 2) (N=79) | BP-CML Total (Part 2) (N=64) | Bosutinib 500 mg, Ph+ ALL (Part 2) (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 2 | 0 | 1 | 1 | 0 | 4 | 5 | 1
Chest pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Asthenia (General disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 4 | 3 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Submandibular mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 6 | 5 | 0 | 0 | 0 | 0 | 9 | 5 | 3
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 2 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis post varicella (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0 | 3 | 3 | 1 | 5 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 | 2 | 0 | 4 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Circumoral oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allogenic bone marrow transplantation therapy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adhesion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perforation bile duct (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneunomia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedure infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bone fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pregnancy of partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Knee anthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Necrosis ischaemic (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 500 mg, CP2L-CML IM-R (Part 2) (N=195) | Bosutinib 500 mg, CP2L-CML IM-I (Part 2) (N=89) | Bosutinib 500 mg, CP3L-CML IM R/I, (D+NI) R/I or NI-I (Part 2) (N=5) | Bosutinib 500 mg, CP3L-CML IM R/I + D-R (Part 2) (N=38) | Bosutinib 500 mg, CP3L-CML IM R/I + D-I (Part 2) (N=50) | Bosutinib 500 mg, CP3L-CML IM R/I + NI-R (Part 2) (N=26) | AP-CML Total (Part 2) (N=79) | BP-CML Total (Part 2) (N=64) | Bosutinib 500 mg, Ph+ ALL (Part 2) (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 61 | 32 | 3 | 9 | 18 | 12 | 35 | 18 | 5
Anaemia (Blood and lymphatic system disorders) | 45 | 24 | 2 | 7 | 7 | 6 | 33 | 19 | 10
Neutropenia (Blood and lymphatic system disorders) | 26 | 13 | 1 | 8 | 6 | 7 | 12 | 16 | 2
Leukopenia (Blood and lymphatic system disorders) | 19 | 8 | 0 | 4 | 1 | 0 | 7 | 9 | 2
Leukocytosis (Blood and lymphatic system disorders) | 7 | 0 | 0 | 1 | 2 | 0 | 4 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 166 | 76 | 5 | 30 | 42 | 22 | 67 | 41 | 15
Nausea (Gastrointestinal disorders) | 85 | 46 | 2 | 20 | 23 | 12 | 36 | 30 | 12
Vomiting (Gastrointestinal disorders) | 73 | 32 | 0 | 14 | 24 | 7 | 35 | 26 | 11
Abdominal pain (Gastrointestinal disorders) | 50 | 24 | 0 | 8 | 12 | 8 | 19 | 11 | 3
Abdominal pain upper (Gastrointestinal disorders) | 41 | 17 | 0 | 8 | 9 | 4 | 9 | 7 | 0
Constipation (Gastrointestinal disorders) | 22 | 17 | 2 | 2 | 7 | 3 | 14 | 9 | 4
Dyspepsia (Gastrointestinal disorders) | 21 | 7 | 0 | 7 | 4 | 1 | 9 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 17 | 8 | 0 | 2 | 4 | 3 | 1 | 4 | 0
Flatulence (Gastrointestinal disorders) | 4 | 6 | 0 | 3 | 3 | 1 | 2 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 8 | 9 | 0 | 1 | 0 | 0 | 4 | 1 | 2
Pyrexia (General disorders) | 58 | 17 | 1 | 5 | 7 | 3 | 28 | 22 | 10
Fatigue (General disorders) | 49 | 24 | 3 | 8 | 12 | 2 | 17 | 13 | 5
Asthenia (General disorders) | 25 | 16 | 2 | 2 | 1 | 4 | 11 | 3 | 5
Oedema peripheral (General disorders) | 17 | 11 | 1 | 1 | 4 | 4 | 6 | 7 | 5
Pain (General disorders) | 16 | 5 | 2 | 2 | 2 | 1 | 6 | 3 | 2
Chest pain (General disorders) | 13 | 7 | 1 | 1 | 2 | 0 | 6 | 3 | 2
Oedema (General disorders) | 9 | 4 | 0 | 2 | 2 | 0 | 5 | 2 | 2
Chills (General disorders) | 13 | 5 | 0 | 0 | 3 | 0 | 3 | 2 | 3
Nasopharyngitis (Infections and infestations) | 25 | 13 | 1 | 3 | 5 | 4 | 7 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 9 | 2 | 3 | 7 | 0 | 8 | 2 | 0
Influenza (Infections and infestations) | 21 | 6 | 1 | 4 | 4 | 3 | 5 | 0 | 1
Urinary tract infection (Infections and infestations) | 20 | 8 | 1 | 1 | 2 | 2 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 42 | 21 | 1 | 6 | 6 | 5 | 11 | 4 | 2
Platelet count decreased (Investigations) | 16 | 11 | 0 | 1 | 1 | 2 | 5 | 4 | 2
Weight decreased (Investigations) | 27 | 8 | 0 | 0 | 7 | 0 | 6 | 3 | 0
Blood creatinine increased (Investigations) | 18 | 8 | 1 | 4 | 6 | 4 | 6 | 3 | 0
Lipase increased (Investigations) | 17 | 9 | 0 | 3 | 2 | 2 | 6 | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 3 | 0 | 3 | 0 | 3 | 5 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 29 | 12 | 1 | 3 | 7 | 4 | 7 | 12 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 5 | 0 | 0 | 3 | 2 | 2 | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 0 | 1 | 0 | 1 | 1 | 5 | 3 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 6 | 1 | 1 | 5 | 0 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 17 | 0 | 5 | 10 | 6 | 12 | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 16 | 1 | 5 | 5 | 3 | 8 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 4 | 0 | 2 | 5 | 3 | 9 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 7 | 0 | 3 | 1 | 1 | 7 | 6 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 3 | 0 | 3 | 5 | 1 | 1 | 7 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0 | 5 | 3 | 2 | 5 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 7 | 0 | 2 | 5 | 1 | 4 | 1 | 2
Headache (Nervous system disorders) | 35 | 18 | 1 | 7 | 15 | 8 | 12 | 13 | 6
Dizziness (Nervous system disorders) | 16 | 9 | 2 | 5 | 8 | 3 | 11 | 7 | 2
Insomnia (Psychiatric disorders) | 6 | 3 | 3 | 1 | 5 | 1 | 8 | 5 | 2
Anxiety (Psychiatric disorders) | 8 | 7 | 0 | 1 | 2 | 1 | 8 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 19 | 2 | 7 | 12 | 4 | 24 | 8 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 9 | 1 | 2 | 9 | 1 | 14 | 12 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 10 | 1 | 2 | 3 | 2 | 8 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 7 | 1 | 3 | 13 | 1 | 8 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 63 | 36 | 2 | 10 | 18 | 3 | 27 | 20 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 9 | 0 | 9 | 8 | 3 | 6 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 16 | 4 | 0 | 1 | 4 | 3 | 3 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 10 | 4 | 0 | 2 | 2 | 2 | 4 | 1 | 0
Hypertension (Vascular disorders) | 17 | 6 | 0 | 2 | 5 | 1 | 6 | 2 | 2
Pericardial effusion (Cardiac disorders) | 3 | 2 | 1 | 1 | 4 | 0 | 4 | 1 | 0
Toothache (Gastrointestinal disorders) | 12 | 6 | 1 | 2 | 2 | 0 | 3 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 1 | 1 | 0 | 1 | 0 | 2 | 5 | 1
Bronchitis (Infections and infestations) | 13 | 3 | 1 | 1 | 2 | 1 | 6 | 0 | 0
Sinusitis (Infections and infestations) | 7 | 3 | 1 | 2 | 4 | 0 | 1 | 1 | 0
Amylase increased (Investigations) | 12 | 3 | 0 | 2 | 1 | 3 | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 38 | 18 | 0 | 2 | 3 | 4 | 12 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 14 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 6 | 10 | 0 | 1 | 0 | 3 | 2 | 0 | 0
Weight increased (Investigations) | 12 | 3 | 0 | 3 | 1 | 0 | 2 | 3 | 0
White blood cell count decreased (Investigations) | 6 | 9 | 0 | 0 | 0 | 0 | 3 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 1
Hypoaesthesia (Nervous system disorders) | 11 | 2 | 0 | 0 | 1 | 1 | 3 | 2 | 1
Paraesthesia (Nervous system disorders) | 11 | 3 | 1 | 0 | 3 | 0 | 2 | 1 | 0
Depression (Psychiatric disorders) | 9 | 4 | 1 | 0 | 3 | 2 | 2 | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 1 | 1 | 5 | 0 | 3 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 2 | 3 | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 3 | 1 | 0 | 3 | 0 | 1 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 3 | 1 | 2 | 0 | 0
Flushing (Vascular disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 0
Eye oedema (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 5 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 7 | 2 | 0 | 1 | 0 | 3 | 4 | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 6 | 3 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 2
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 2 | 0 | 0 | 2 | 1 | 4 | 1 | 0
Face oedema (General disorders) | 4 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Influenza like illness (General disorders) | 6 | 5 | 1 | 1 | 3 | 0 | 1 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 4 | 2 | 0
Oral herpes (Infections and infestations) | 3 | 3 | 0 | 1 | 0 | 1 | 6 | 1 | 0
Pharyngitis (Infections and infestations) | 6 | 5 | 1 | 2 | 0 | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 1 | 3 | 1 | 2 | 4 | 1
Respiratory tract infection viral (Infections and infestations) | 4 | 3 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Blood urea increased (Investigations) | 3 | 1 | 0 | 2 | 2 | 0 | 2 | 1 | 0
Blood uric acid increased (Investigations) | 11 | 1 | 0 | 2 | 2 | 0 | 4 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 2 | 0 | 3 | 0 | 1 | 2 | 0 | 0
Globulins decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 5 | 0 | 0 | 1 | 0 | 3 | 1 | 2
White blood cells urine positive (Investigations) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 2 | 0 | 2 | 1 | 2 | 4 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 2 | 0 | 0 | 1 | 4 | 4 | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 1 | 0 | 2 | 4 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 1 | 0 | 3 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0 | 0 | 2 | 1 | 4 | 0
Dysgeusia (Nervous system disorders) | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 3 | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Syncope (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 6 | 4 | 0 | 3 | 0 | 2 | 1 | 2 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 1 | 0 | 1 | 1 | 0 | 5 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 5 | 0 | 0 | 2 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 7 | 0 | 1 | 2 | 2 | 4 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 1 | 3 | 1 | 2 | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 3
Skin burning sensation (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 7 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 5 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Analyses of progression free survival and overall survival was based on all-treated population, instead of evaluable population which was the primary efficacy population as per planned analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.